CLINICAL TRIAL: NCT01865578
Title: Transcranial Direct Current Stimulation on Cortical Plasticity in Patients With Anti-NMDA Receptor Encephalitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Agnes Flöel, Prof. Dr. med Agnes Floeel, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EA1/037/12
Record Dates: First submitted 2013-05-21; First posted 2013-05-31 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Anti-NMDA Receptor Encephalitis
MeSH Terms: conditions — Anti-N-Methyl-D-Aspartate Receptor Encephalitis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- tDCS (Experimental): Transcranial direct current stimulation
  Interventions: Device: tDCS
- sham stimulation (Sham Comparator): sham stimulation
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: tDCS — Transcranial direct current stimulation involves the application of weak electric currents to the brain.
  Arms: tDCS
Device: Sham Stimulation — no electrical stimulation
  Arms: sham stimulation

SUMMARY:
Patients suffering from anti-NMDA receptor encephalitis show impaired NMDA-receptor dependent neuronal transmission. Furthermore, they often have cognitive deficits of different magnitude. Impaired neuronal signaling of NMDA-receptors very likely result in decreased cortical synaptic plasticity. Thus, this represents one major reason of cognitive deficits. Synaptic plasticity can be assessed in humans via the non-invasive technique of transcranial magnetic stimulation (TMS).

The current study aims to investigate whether learning ability and also cortical plasticity can be changed by applying sessions of transcranial direct current stimulation (tDCS). Therefore, we are recruiting 10 to 15 patients suffering from anti-NMDA receptor encephalitis as well as healthy controls in order to compare tDCS effects. Learning ability is assessed by motor sequence tasks, whereas cortical plasticity is measured via TMS.

tDCS is a novel non-invasive technique allowing induction of changes in cerebral excitability level and also cortical plasticity. Previous studies showed positive outcome of anodal stimulation on learning tasks. Especially motor learning seems to be an important target for tDCS treatment since it showed best results for both post-stroke patients and healthy subjects. Multiple sessions of tDCS are inducing long-term effects and improved learning function, which were present three months after stimulation.

In this study we hope to reveals new insights into the pathomechanisms of impaired cognitive and learning abilities in patients having anti-NMDA receptor encephalitis. Moreover, we evaluate whether tDCS is an effective treatment for patients with cognitive and learning deficits.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from anti-NMDA receptor encephalitis
* healthy (control) subjects

Exclusion Criteria:

* Any metal inside the body/head, e.g. clips, pace maker, medical pumps, cochlear implant etc.
* Traumatic brain injury
* Stroke
* Cerebral tumor
* Pregnancy
* untreated severe internal or psychiatric diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
neurophysiological measurements using TMS | 1 week
  TMS protocoll (a paired associative stimulation) is applied after tDCS or sham stimulation

SECONDARY OUTCOMES:
performance in a motor task | 1 week
  performance in a motor task is compared after a tDCS or sham stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Floeel, Prof. MD, Principal Investigator — Charite University
Locations (1):
- Charite University Medicine, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Volz MS, Finke C, Harms L, Jurek B, Paul F, Floel A, Pruss H. Altered paired associative stimulation-induced plasticity in NMDAR encephalitis. Ann Clin Transl Neurol. 2016 Jan 16;3(2):101-13. doi: 10.1002/acn3.277. eCollection 2016 Feb. PMID 26900584